CLINICAL TRIAL: NCT00366015
Title: Same Procedure Cardiac Hybrid Surgery in a Specialty Built OR-- A Pilot Study
Brief Title: Coronary Stenting and Coronary Bypass Grafting at the Same Time in a Specialty Built Operating Room
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Canada Foundation for Innovation (Other); Ontario Innovative Trust (Unknown); Ontario Research and Development Challenge Fund (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R-04-158; 9874 (Other: REB)
Record Dates: First submitted 2006-08-16; First posted 2006-08-18 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; PCI; Drug eluting stents; Coronary Hybrid Revascularization; Robotic CABG
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Robotic-assisted Coronary Surgical Revascularization — Robotic assistance of coronary artery bypass grafting using the DaVinci surgical robotic console
Procedure: PCI- Drug Eluting Stents — Drug eluting stents performed by cardiologist within the same operating theatre following robotic assisted coronary artery bypass surgery

SUMMARY:
This study will combine coronary stenting with minimally invasive robotic coronary bypass surgery, accomplished with the use of the da Vinci robot, to restore blood flow to occluded coronary arteries. Two previously approved and commonly performed procedures used to treat coronary artery disease(coronary stenting and robotic bypass surgery) are being combined into a hybrid surgery in a specialty built operating room. Patients with low risk coronary lesions will undergo cardiac hybrid revascularization using stenting and LIMA to LAD robotic bypass concomitantly. Patients' postoperative bleeding rates, angiographs and complication free rates will be recorded.

DETAILED DESCRIPTION:
Coronary artery disease (CAD) is the leading cause of death in the United States and becomes more common as the population ages (American Heart Association, 2003). The symptoms of CAD may not become perceptible until the condition has advanced to a severe and serious stage, which might explain the large mortality and morbidity rates associated with heart disease.

At this point there are many procedures available to treat CAD all of which aim to improve myocardial blood flow, stop angina, increase exercise ability and ultimately free patients from medications and improve their quality of life. Medications are used to reduce blood pressure and relieve strain on the heart. Cardiologists use angioplasty, which compresses plaque deposits, and stenting, in which a small wire mesh tube is inserted into the diseased artery to revascularize the heart muscle. On-pump coronary artery bypass grafting (CABG) redirects blood flow around clogged vessels of the heart and is commonly used by cardiac surgeons to treat CAD because it has been proven to yield the lowest restenosis rate of all revascularization techniques (Cisowski, 2002). CABG is an effective yet painful and traumatic intervention.

The desire to discover a less distressing approach to coronary artery revascularization has led to a fairly new cardiac hybrid procedure that involves stenting followed by a minimally invasive left internal mammary artery (LIMA) to left anterior descending artery (LAD) bypass graft (Amodeo, 2002). The hybrid procedure for revascularization carries a lower morbidity than does on-pump CABG and is also quickly gaining acceptance in the surgical community (de Canniere et al, 2001). The two procedures of hybrid revascularization are currently performed within 24 to 48 hours of each other with little collaboration between cardiac surgeons and cardiologist.

This study will asses the efficacy and safety of cardiac hybrid surgery that combines stenting and robotic LIMA to LAD grafting in the same procedure in a specialty built operating room. Long term use of the antiplatelet inhibitor, clopidogrel, to be taken by patients in this study, was proven to significantly reduce the risk of adverse ischemic events after percutaneous coronary interventions (Steinhubl, 2002). In addition, the application of Bivalirudin (Direct Thrombin Inhibitor) will be assessed in this integrated myocardial revascularization scenario. The many attractive aspects of robotic hybrid bypass include the avoidance of the procedural phases (arrested heart, blood transfusion, median sternotomy and cardiopulmonary bypass) of on-pump CABG. Robotic LIMA to LAD bypass and stenting in the same procedure will allow cardiac surgeons and cardiologists to work together to help patients obtain safe and effective coronary artery revascularization.

ELIGIBILITY:
Inclusion Criteria:

* Patients with class A or B1 low risk coronary artery lesion as defined by TIMI

Exclusion Criteria:

* Contraindications to PCI which include:

Occluded coronary vessels, PVD, Unable to achieve access, Fresh thrombus, Vessels <1.5mm

* Contraindications to Robotic Surgery which include:

Buried LAD, Unable to tolerate single lung ventilation, Inability to undergo beating heart surgery, Previous surgery of the left chest cavity, Lack of intrathoracic work space, Patients requiring emergency surgery,

The following patients are also excluded:

Patients with coagulation disorders; inability to tolerate GIIb/III inhibitors, Patients with ventricular arrhythmias, Patients with severe non-cardiac conditions with poor prognosis, Patients with a BMI >40, Patients with an ejection fraction of <30%, Patients with chronic renal insufficiency and creatinine >200umol/L, Patients who are >85 years of age, Patients participating in any other investigational device or study drug, Patients who have had previous thoracic surgery, Patients who have a pre-op intra-aortic balloon pump, Patients who are not able to follow the protocol requirements, Patients undergoing concomitant surgery; CABG + Valve surgery

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2003-07-29 (Actual); Primary Completion 2010-12-31 (Actual); Study Completion 2010-12-31 (Actual)

PRIMARY OUTCOMES:
Safety & efficacy of integrated myocardial revascularization performed in a single stage | 5 years post end of study

SECONDARY OUTCOMES:
One-year postoperative stenosis rate (Stenosis may be evaluated by the angiographic documentation of blood flow). | One year
Success rate is defined as a reduction in stenosis to < 50%. | One year
Myocardial infarction, | within 30 days of surgery
Death, | within 30 days of surgery and/or within primary hospitalization
Repeat revascularization at any time after the robotic hybrid revascularization (Repeat revascularization are those involving a previously treated lesionfollowing the initial hybrid procedure) | One year
In-hospital complications during or after surgery, | within initial hospitalization or within 30 days of discharge
Inability to revascularize with the use of both stenting and LIMA to LAD bypass, | within initial hospitalization
Inability to revascularize with the use of the da Vinci Surgical System | within initial hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Bob Kiaii, MD, FRCSC, Principal Investigator — Department of Cardiac Surgery, University of Western Ontario and the London Health Sciences Centre, University Hospital
Locations (1):
- The London Health Sciences Centre, University Hospital, London, Ontario, Canada

REFERENCES:
- [Background] Merry AF, Raudkivi PJ, Middleton NG, McDougall JM, Nand P, Mills BP, Webber BJ, Frampton CM, White HD. Bivalirudin versus heparin and protamine in off-pump coronary artery bypass surgery. Ann Thorac Surg. 2004 Mar;77(3):925-31; discussion 931. doi: 10.1016/j.athoracsur.2003.09.061. PMID 14992900
- [Background] Koster A, Spiess B, Chew DP, Krabatsch T, Tambeur L, DeAnda A, Hetzer R, Kuppe H, Smedira NG, Lincoff AM. Effectiveness of bivalirudin as a replacement for heparin during cardiopulmonary bypass in patients undergoing coronary artery bypass grafting. Am J Cardiol. 2004 Feb 1;93(3):356-9. doi: 10.1016/j.amjcard.2003.10.021. PMID 14759391
- [Background] Vassiliades TA Jr, Douglas JS, Morris DC, Block PC, Ghazzal Z, Rab ST, Cates CU. Integrated coronary revascularization with drug-eluting stents: immediate and seven-month outcome. J Thorac Cardiovasc Surg. 2006 May;131(5):956-62. doi: 10.1016/j.jtcvs.2005.10.058. Epub 2006 Apr 27. PMID 16678575
- [Background] Katz MR, Van Praet F, de Canniere D, Murphy D, Siwek L, Seshadri-Kreaden U, Friedrich G, Bonatti J. Integrated coronary revascularization: percutaneous coronary intervention plus robotic totally endoscopic coronary artery bypass. Circulation. 2006 Jul 4;114(1 Suppl):I473-6. doi: 10.1161/CIRCULATIONAHA.105.001537. PMID 16820621
- [Background] Cisowski M, Morawski W, Drzewiecki J, Kruczak W, Toczek K, Bis J, Bochenek A. Integrated minimally invasive direct coronary artery bypass grafting and angioplasty for coronary artery revascularization. Eur J Cardiothorac Surg. 2002 Aug;22(2):261-5. doi: 10.1016/s1010-7940(02)00262-2. PMID 12142196
- [Background] Zenati M, Cohen HA, Griffith BP. Alternative approach to multivessel coronary disease with integrated coronary revascularization. J Thorac Cardiovasc Surg. 1999 Mar;117(3):439-44; discussion 444-6. doi: 10.1016/s0022-5223(99)70322-3. PMID 10047645
- [Background] Angelini GD, Wilde P, Salerno TA, Bosco G, Calafiore AM. Integrated left small thoracotomy and angioplasty for multivessel coronary artery revascularisation. Lancet. 1996 Mar 16;347(9003):757-8. doi: 10.1016/s0140-6736(96)90107-5. No abstract available. PMID 8602013
- [Background] Bonatti J, Schachner T, Bonaros N, Laufer G, Kolbitsch C, Margreiter J, Jonetzko P, Pachinger O, Friedrich G. Robotic totally endoscopic coronary artery bypass and catheter based coronary intervention in one operative session. Ann Thorac Surg. 2005 Jun;79(6):2138-41. doi: 10.1016/j.athoracsur.2003.12.074. PMID 15919329
- [Background] Bonatti J, Schachner T, Bonaros N, Jonetzko P, Ohlinger A, Lockinger A, Stalzer B, Eschertzhuber S, Friedrich G. Treatment of double vessel coronary artery disease by totally endoscopic bypass surgery and drug-eluting stent placement in one simultaneous hybrid session. Heart Surg Forum. 2005;8(4):E284-6. doi: 10.1532/HSF98.20051136. PMID 16112943
- [Background] Dogan S, Aybek T, Andressen E, Byhahn C, Mierdl S, Westphal K, Matheis G, Moritz A, Wimmer-Greinecker G. Totally endoscopic coronary artery bypass grafting on cardiopulmonary bypass with robotically enhanced telemanipulation: report of forty-five cases. J Thorac Cardiovasc Surg. 2002 Jun;123(6):1125-31. doi: 10.1067/mtc.2002.121305. PMID 12063459